CLINICAL TRIAL: NCT01941615
Title: An Open-label, Two-period, Fixed-sequence, Phase I Trial to Evaluate the Effect of Multiple Doses of BI 207127 + Faldaprevir on the Multiple-dose Pharmacokinetics of a Combination of Ethinylestradiol and Levonorgestrel in Healthy Premenopausal Female Subjects
Brief Title: Effect of BI 207127 + Faldaprevir on Blood Levels of Oral Contraceptives Containing Ethinylestradiol and Levonorgestrel
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1241.31; 2013-000298-62 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
MeSH Terms: interventions — faldaprevir; ethinyl estradiol, levonorgestrel drug combination; deleobuvir

ARMS (1):
- BI 207127 + faldaprevir + Microgynon (Experimental): Period A: Microgynon®; Period B: Microgynon® + FDV + BI 207127
  Interventions: Drug: faldaprevir; Drug: Microgynon®; Drug: BI 207127

INTERVENTIONS:
Drug: faldaprevir — oral doses for 10 days (period B)
Drug: Microgynon® — oral doses for 23 days (period A+B)
Drug: BI 207127 — oral doses for 10 days (period B)

SUMMARY:
Investigate the effect of multiple oral doses of BI 207127 + faldaprevir (FDV) on the multiple dose pharmacokinetics of ethinylestradiol and levonorgestrel (Microgynon®) in healthy premenopausal female volunteers.

ELIGIBILITY:
Inclusion criteria:

* Healthy female subjects
* Age 18 to 35 years (inclusive)
* Body Mass Index 20-29.9 kg/m2
* Use of hormonal contraception (i.e. oral contraceptives, hormonal contraceptive vaginal ring, but not hormone-containing intrauterine devices, depot injections or contraceptive implants)

Exclusion criteria:

* Any relevant deviation from healthy conditions
* Subject is assessed by the investigator as unsuitable for inclusion, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Positive pregnancy test, pregnancy or planning to become pregnant within 1 month of study completion, or lactation
* Any relevant finding of the gynaecological examination
* Thrombotic predisposition according to thrombophilic testing
* Existing or history of arterial thrombotic or embolic processes, conditions which predispose to them e.g. disorders of the clotting processes, valvular heart disease and atrial fibrillation
* Existing or history of confirmed venous thromboembolism, family history of venous thromboembolism, and other known risk factors for venous thromboembolism.
* Relevant varicosis
* No use of an additional contraceptive method from screening examination until 1 month after last study drug administration (acceptable methods are considered to be barrier methods, sexual abstinence, non-hormone-containing intrauterine device, or vasectomisation for the male partner).

Use of hormone-containing intrauterine device, depot injection or contraceptive implants

* Any history of relevant liver diseases (e.g. disturbances of liver function, jaundice or persistent itching during a previous pregnancy, Dubin-Johnson syndrome, Rotor syndrome, or previous or existing liver tumours)
* AST (aspartate transaminase) and/or ALT (alanine transaminase) > 1.5 ULN (upper limit of normal)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1241.31.2 Boehringer Ingelheim Investigational Site, Mannheim, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was planned to include 18 healthy premenopausal female subjects. Because this trial was prematurely discontinued during the run-in period, only 16 subjects were entered.
Groups:
- Deleobuvir + Faldaprevir + Microgynon: This was an open-label, 2-period, fixed-sequence study. After a run-in period of 28 to 56 days (treatment with Microgynon® once daily for 21 to 49 days, depending on the menstrual cycle, followed by a tablet-free interval of 7 days), subjects were to begin the first (reference) treatment period of Microgynon® alone for 13 days, immediately (without washout) followed by the second (test) treatment period of Microgynon® plus deleobuvir+faldaprevir for 10 days.
Period: Run in Treatment: Microgynon®
Arm/Group | Deleobuvir + Faldaprevir + Microgynon
Started | 16
Completed | 16
Not Completed | 0
Period: Reference Treatment: Microgynon®
Arm/Group | Deleobuvir + Faldaprevir + Microgynon
Started | 0
Completed | 0
Not Completed | 0
Period: Microgynon® Plus Deleobuvir+Faldaprevir
Arm/Group | Deleobuvir + Faldaprevir + Microgynon
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Deleobuvir + Faldaprevir + Microgynon
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: AUCtau,ss of Ethinylestradiol
Description: Area under the concentration-time curve of ethinylestradiol in plasma at steady state over a uniform dosing interval t (AUCtau,ss).
Time Frame: Visit (V)3: 2 hours(h) pre dose, 240, 264, 288, 288.5, 289, 289.5, 290, 291, 292, 294, 296, 298, 300 h post dose; V4: 0, 24, 48, 72, 96, 120, 144, 168, 192, 216, 216.5, 217, 217.5, 218, 219, 220, 222, 224, 226, 228, 240 h post dose for oral contraceptives
Population: Since this trial was prematurely discontinued during the run-in period, no blood samples for pharmacokinetics were collected and therefore no pharmacokinetic endpoints could be determined.
Arm/Group | Deleobuvir + Faldaprevir + Microgynon
Number analyzed (Participants) | 0

2. Primary Outcome: Cmax,ss of Ethinylestradiol
Description: Maximum measured concentration of ethinylestradiol in plasma at steady state over a uniform dosing interval t
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Deleobuvir + Faldaprevir + Microgynon
Number analyzed (Participants) | 0

3. Primary Outcome: C24,ss of Ethinylestradiol
Description: Measured concentration of ethinylestradiol in plasma at steady state 24 hours after drug administration.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Deleobuvir + Faldaprevir + Microgynon
Number analyzed (Participants) | 0

4. Primary Outcome: AUCtau,ss of Levonogestrel
Description: Area under the concentration-time curve of levonogestrel in plasma at steady state over a uniform dosing interval t.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Deleobuvir + Faldaprevir + Microgynon
Number analyzed (Participants) | 0

5. Primary Outcome: Cmax,ss of Levonogestrel
Description: Maximum measured concentration of levonogestrel in plasma at steady state over a uniform dosing interval t.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Deleobuvir + Faldaprevir + Microgynon
Number analyzed (Participants) | 0

6. Primary Outcome: C24,ss of Levonogestrel
Description: Measured concentration of levonogestrel in plasma at steady state 24 hours after drug administration.
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Deleobuvir + Faldaprevir + Microgynon
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: until end of run-in period up to 49 days
Description: study was terminated after run-in period
Groups:
- Deleobuvir + Faldaprevir + Microgynon: In the run-in period starting between Day -56 and Day -28, all subjects were to take 1 Microgynon® tablet (combined oral contraceptive ethinylestradiol / levonorgestrel) once daily for 21 to 49 days (depending on the menstrual cycle) until Day -8.
  In the last 7 days of the run-in period (Day -7 to Day -1), no treatment was given in order to induce withdrawal bleeding. The next day was to be Day 1 of the study. Subjects who were using oral contraceptives before the study started the run-in period after the usual tablet-free interval of 7 days.
  Subjects who were using hormonal contraceptive vaginal rings before the study started the run-in-period after the usual hormone-free interval of 7 days.
Arm/Group | Deleobuvir + Faldaprevir + Microgynon
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 4/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deleobuvir + Faldaprevir + Microgynon (N=16)
Nasopharyngitis (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 2
Uterine pain (Reproductive system and breast disorders) | 1

LIMITATIONS AND CAVEATS:
This trial was prematurely discontinued during the run-in period. During the run-in period, subjects were to receive Microgynon® once daily for 21 to 49 days. The investigational products Deleobuvir + faldaprevir were not administered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.